CLINICAL TRIAL: NCT03426462
Title: Time to Peak Effect of Propofol in Children
Acronym: TPEPC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UKBB-2017/032
Record Dates: First submitted 2018-01-25; First posted 2018-02-08 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Propofol; Child
Keywords: Pharmacodynamic; Permutation Entropy; EEG
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Intervention Model Description: Age groups 1-6 years will be compared with 8-13 years whilst undergoing propofol anesthesia to detect whether there is indeed a difference in the speed of onset of the hypnotic effect of the drug.
Who Masked: Outcomes Assessor
Masking Description: The analysis of the electroencephalogram will be blinded to the age of the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Age 1-6 years (Experimental): Induction of anesthesia with propofol using infusion pumps that are programmed with a pharmacokinetic model to achieve a calculated plasma concentration of the drug; this is followed by two anesthetic deepening episodes.
  The target plasma concentrations achieved, as calculated by the programmed pump, is exactly the same in both age groups.
  Interventions: Drug: Propofol
- Age 8-13 years (Experimental): Induction of anesthesia with propofol using infusion pumps that are programmed with a pharmacokinetic model to achieve a calculated plasma concentration of the drug; this is followed by two anesthetic deepening episodes.
  The target plasma concentrations achieved, as calculated by the programmed pump, is exactly the same in both age groups.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Induction of anesthesia and two further deepening episodes will be performed whilst recording the electroencephalogram.

SUMMARY:
In order to determine the speed of onset of the anaesthetic propofol in children, investigators will compare the two age groups 1-6 years vs 8-13 years. The primary outcome measure is the time to peak effect of a bolus of proposal, which is measured by analysing the electroencephalogram by using the permutation entropy. Further pharmacodynamic modelling will enable investigators to quantify the difference with age in the hypnotic effect of propofol.

ELIGIBILITY:
Inclusion Criteria:

* The study population will be healthy children in the ranges of 1-6 and 8-13 years of age having surgery with American Society of Anaesthesia (ASA) grades I-II (ie. no prior functional limitation due to comorbidities) that fulfil the following points:
* parental written consent obtained at least a day prior to begin of the subject's study episode; and
* the child is appropriate for induction and maintenance of anaesthesia with propofol.

Exclusion Criteria:

* Any significant subject co-morbidity (ASA III or IV);
* Withdrawal of consent/assent at any point in the study;
* Failure to cannulate a peripheral vein prior to induction after two attempts;
* Any other reason making IV induction with propofol impossible;
* Allergy to propofol (or its emulsion carrier), Eutectic Mixture of Local Anesthetics (EMLA) cream or Nitrous Oxide (N2O);
* previous enrolment in the study;
* Any anaesthetic problem that would take precedence over completion of the study protocol.

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Time to peak effect of a propofol bolus | up to 20 minutes from baseline until peak effect following second bolus administration
  This is the time from the start of the propofol bolus administration to the maximal suppression of the electroencephalogram; per subject two boli will be administered

CONTACTS AND LOCATIONS:
Overall Officials: Gil Gavel, Principal Investigator — Universitäts Kinderspital beider Basel (UKBB)
Locations (1):
- Universitäts Kinderspital beider Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No